CLINICAL TRIAL: NCT05976256
Title: Kinesiotaping in Trauma
Acronym: KIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: OLVG (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WO 21.210
Record Dates: First submitted 2023-07-17; First posted 2023-08-04 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Fracture Rib; Acromioclavicular Joint Dislocation; Fracture Clavicle; Fracture, Proximal Humeral
Keywords: kinesiotaping
MeSH Terms: conditions — Rib Fractures; Shoulder Fractures

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Kinesiotape (Active Comparator): Patients receives the additional treatment with kinesiotaping (and also standard treament)
  Interventions: Other: sham tape (leukotape classic); Other: standard treatment
- sham tape (Sham Comparator): patient receives an additional treatment with sham tape (without elastic features) (and also standard treatment)
  Interventions: Other: Kinesio taping; Other: standard treatment
- control group (No Intervention): patient receives the standard treamtment without additional tape treatment

INTERVENTIONS:
Other: Kinesio taping — Kinesio tape is a thin, elastic tape that applies pressure to the skin (because of the elasticity of the tape), reducing pain by reducing nociceptive stimulation.
  Other Names: Leukotape K; medical taping
  Arms: sham tape
Other: sham tape (leukotape classic) — leuko tape classic is used in this study to explore the possible placebo effect of kinesiotape
  Other Names: non elastic tape
  Arms: Kinesiotape
Other: standard treatment — standard treatment is the treatment with oral analgesics and a sling (if shoulder injury)
  Arms: Kinesiotape; sham tape

SUMMARY:
Rationale: Patients with acute traumatic injury to the shoulder or chest wall in de Emergency Department (ED) usually have intense pain. The patient normally is treated with oral analgesics as standard care and in shoulder injury with a sling. Pain of the shoulder or chest wall increases with movement of the affected arm and chest. Kinesiotaping is offered regularly as an additional pain treatment, but there is no hard evidence about its effectiveness. A randomized pilot study in OLVG (Bakker 2022) showed the pain decreasing more when using kinesiotaping comparing to no tape. However, a placebo-effect could not be ruled out and the pilot data need confirmation in a large cohort of patients to study the effectiveness of additional treatment with kinesiotaping in terms of pain, comfort and patient satisfaction.

DETAILED DESCRIPTION:
Objective: The primary aim of this study is to evaluate the effect of kinesiotaping on number of patients with clinically meaningful pain reduction after 1 week in patients with acute traumatic injury in shoulder or chest wall, compared to sham tape and no tape. The secondary aims are to assess the effect of kinesiotaping on pain reduction at 15 min, 3 weeks and 8 weeks, and the effects on the skin, use of oral analgesics, independence, activity pattern, progress of pain symptoms, comfort and patient satisfaction at 1, 3 and 8 weeks. Also the need of physiotherapy is one of the secondary aims.

Study design: Parallel randomized controlled trial with three arms

Study population: Patients of or over 18 years old with an acute single shoulder or chest wall injury (rib fracture, disruption of the acromioclavicular (AC) joint Tossy type 1 and 2, not or hardly dislocated fracture of clavicle or proximal humeral bone).

Intervention (if applicable): One group will receive treatment with kinesiotaping, another group receives sham taping (no elastic tape) and the third group receives no taping. This treatment is additional to the general treatment with oral analgesics and a sling (when shoulder injury).

Main study parameters/endpoints: The main study parameter is the proportion of patients who experienced a clinically meaningful reduction in pain score (≥2 points on NRS) at week 1 compared to T1. The kinesiotape group will be compared to the sham group and to the control group.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

At 15 minutes after receiving kinesio tape, sham tape or no tape, 1 week, 3 weeks and 8 weeks after visiting the emergency department the pain of these patients is evaluated using NRS by the Brief Pain Inventory (BPI). The effect of use of oral analgesics (questionnaire), on the skin (questionnaire), on independence, activity pattern and progress of pain symptoms (Groningen Activity Restriction Scale (GARS)), comfort and patient satisfaction (Global Perceived Effect (GPE-DV)) is evaluated after 1, 3 and 8 weeks. Physiotherapy is elevated after 8 weeks. Due to the limited seriousness of the injury and the non-invasive nature of the interventions, any serious complication or adverse event is not expected. Benefits of participating this study could be pain reduction in the affected body part.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Acute injury (occurred <24 hours ago)
* Single shoulder or chest wall injury, which includes one of the following injuries:

  * rib fracture
  * disruption of the AC-joint Tossy type 1 and 2
  * not or hardly dislocated fracture of the clavicle
  * Not or hardly dislocated fracture of the r proximal humeral fracture

Exclusion Criteria:

* • Patients younger than 18 years

  * Incapacitated persons
  * Refusal of participation
  * Intubation indication
  * Decrease of Consciousness
  * Hemodynamic instability
  * 3 or more rib fractures
  * Rib fracture rib 1-3
  * Indication for surgery
  * Hospitalization required
  * Presence of a haemo- or pneumothorax with chest drain indication
  * Already known with allergy for adhesive tape
  * Patients with very thin or loose skin on the applicable body part
  * Skin infection/irritation or open wound on the applicable body part
  * Patients who do not speak Dutch or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
number of patients with clinically meaningful pain reduction | 1 week
  To evaluate the effect of kinesiotaping on number of patients with clinically meaningful pain reduction (Brief Pain Inventory (BPI)) after 1 week in patients with acute traumatic injury in shoulder or chest wall, compared to sham tape and no tape (2 comparisons).

SECONDARY OUTCOMES:
number of patients with clinically meaningful pain reduction | after 15 minutes, 3 weeks and 8 weeks
  the proportion of patients who experience a clinically meaningful reduction in pain score (≥2 points on NRS by BPI). The kinesiotape group will be compared to the sham group and to the control group (2 comparisons).
evaluating skin defects by questionnaire | 1 week, 3 weeks and 8 weeks
  To assess potential skin abnormalities resulting from kinesio taping, a questionnaire will be distributed among the participants. This questionnaire is designed based on the decubitus stages. Additionally, in case of skin abnormalities or rashes, participants will be requested to upload a photograph of the affected area for independent evaluation of the skin condition.
evaluating use of oral analgesics by questionnaire | after 1 week, 3 weeks and 8 weeks
  To evaluate the utilization of oral analgesics, a questionnaire is administered to the participants to ascertain the type of medication employed, as well as to quantify the frequency and dosage of its usage.
evaluating independence, pattern of activity and course of pain complaints by Groningen Activity Restriction Scale (GARS) | after 1 week, 3 weeks and 8 weeks
  To delineate the independence, pattern of activity, and course of pain complaints, we employ the Groningen Activity Restriction Scale (GARS).
Evaluating comfort and patient satisfaction by Global Perceived Effect (GPE-DV) | after 15 minutes, 1 week, 3 weeks and 8 weeks
  To gauge comfort and patient satisfaction, the Global Perceived Effect (GPE-DV) is utilized as a measurement tool.
Evaluating the need of physiotherapy by questionnaire | 8 weeks
  To gain insight into whether patients avail or have availed themselves of physiotherapy, a questionnaire is dispatched after 8 weeks, encompassing queries regarding the utilization of physiotherapy during the treatment period, its frequency, and the nature of the treatment sought.

OTHER OUTCOMES:
clinical meaningful pain reduction for the different intervention arms | 15 min, 1 week, 3 weeks and 8 weeks
  In an exploratory analysis, we would like to assess in a subgroup analysis if the number of patients with clinically meaningful pain reduction after 15 minutes, 1 week, 3 weeks and 8 weeks for the different intervention arms differs between patients with uncomplicated rib fracture, disruption of the AC-joint, clavicle fracture, and proximal humeral fracture (using the BPI-NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Bakker, MSc, Principal Investigator — OLVG; Maro Sandel, MD, PhD, Study Chair — OLVG; Carel Goslings, MD, PhD, Study Chair — OLVG; Janneke Schuitenmaker, MSc, Study Chair — OLVG
Locations (1):
- Mireille Bakker, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No